CLINICAL TRIAL: NCT05112354
Title: Predictive Factors for Recovery in Idiopathic Sensory Neural Hearing Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, suhaib abdelzaker Mohamed, Resident doctor in otolaryngology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Predictive factors in ISSNHL
Record Dates: First submitted 2019-09-24; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Sudden SNHL

STUDY DESIGN:
Intervention Model Description: -If the patient come at first two weeks of onset of hearing loss the patient will be manged by oral corticosteroid in the form of ,prednisolone60mg in two divided doses for 2 weeks.
  2-Patient will be manged by 5 sessions of intratympanic steroid after failure of systemic steroid and patient who come after 2 weeks of onset of hearing loss , each session will be 3 days apart. The injectable material will be 1ml of hydrocortisone 8ml. The injection will be done under local anesthesia and microscope magnification. A pack of lidocaine gel will be applied in the external canal for 10 minutes in EAC to induce anesthesia by using insulin syringe 1ml bore.
  An 8 ml of hydrocortisone will be injected in the ME through posteroinferior part of TM All patients will receive antiviral therapy in the form of acyclovir,valcyclovir All the patient will receive vasodilator.
Masking Description: both the invistigator and care provider donot know the detailes of audiological evalution of the patient nor the comobidities of the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the main group (Experimental): Management plan
  1. If the patient come at first two weeks of onset of hearing loss the patient will be manged by oral corticosteroid in the form of ,prednisolone60mg in two divided doses for 2 weeks.
  2. Patient will be manged by 5 sessions of intratympanic steroid after failure of systemic steroid and patient who come after 2 weeks of onset of hearing loss , each session will be 3 days apart. The injectable material will be 1ml of hydrocortisone 8ml. The injection will be done under local anesthesia and microscope magnification. A pack of lidocaine gel will be applied in the external canal for 10 minutes in EAC to induce anesthesia by using insulin syringe 1ml bore.
  An 8 ml of hydrocortisone will be injected in the ME through posteroinferior part of TM All patients will receive antiviral therapy in the form of acyclovir,valcyclovir All the patient will receive vasodilator
  Interventions: Drug: systemic and intratympanic injection of steoid

INTERVENTIONS:
Drug: systemic and intratympanic injection of steoid — -If the patient come at first two weeks of onset of hearing loss the patient will be manged by oral corticosteroid in the form of ,prednisolone60mg in two divided doses for 2 weeks.
  2-Patient will be manged by 5 sessions of intratympanic steroid after failure of systemic steroid and patient who come after 2 weeks of onset of hearing loss , each session will be 3 days apart. The injectable material will be 1ml of hydrocortisone 8ml. The injection will be done under local anesthesia and microscope magnification. A pack of lidocaine gel will be applied in the external canal for 10 minutes in EAC to induce anesthesia by using insulin syringe 1ml bore.
  An 8 ml of hydrocortisone will be injected in the ME through posteroinferior part of TM All patients will receive antiviral therapy in the form of acyclovir,valcyclovir All the patient will receive vasodilator.
  Other Names: Microscopic Intratympanic steroid injection

SUMMARY:
Sudden sensorineural hearing loss (SSNHL) is an otological emergency that is defined as a hearing loss greater than 30 dB over three consecutive frequencies within 72 hours, with abnormalities of the cochlea, auditory nerve, or central auditory system.1 During 2006 and 2007, the annual incidence of SSNHL was 5-27/100,000 persons per year in the United states.2,3 The causative etiologies for SSNHL included viruses, microcirculation abnormalities, and autoimmune disorders. However, definitive evidence remains elusive.4,5 Currently, steroids are the treatment of choice due to their effects on the inner ear such as immunosuppression and circular enhancement.6,7 Combined systemic and intra-tympanic steroid treatment has previously been reported to be beneficial for SSNHL patients, with overall better treatment outcomes.8,9 However, due to the heterogeneous pathological nature and spontaneous recovery potential of the disease, few controlled studies exist in the literature. As a result, the treatment strategies of SSNHL remain a controversial issue in clinicalpractice .10 The condition exhibits a wide age distribution , with an average of 50-60 years and no sex preference. The hearing loss is unilateral in most Population studies of sudden sensorineural hearing loss cases, with bilateral involvement reported in less than 5%. 11 The severity of the hearing loss is divided roughly equally into mild, moderate, and severe profound. The configuration of the hearing loss varies and can affect high, low, or all frequencies. Tinnitus occurs in about 80% of patients, and vertigo, indicating an associated peripheral vestibular dysfunction, in about 30%. 12 The response to medical therapy shows inconsistent results regarding symptoms especially hearing loss may be due to the uncertainty about the cause of the disease and its progress. little is known about the factors which may contribute to either success or failure of the medical therapy.

Aim of work

1. To evaluate the factors contributing to the success or failure of standardized medical therapy in cases of ISSNHL
2. To detect the degree of correlation of the presenting symptoms and comorbidities to the patient final hearing prognosis.

DETAILED DESCRIPTION:
Patient and methods Study design The study will be conducted as across sectional observation study. Study setting ENT Department Assiut University Hospital outpatient clinic in the period between the 1st July 2019 end of June 2021.

Inclusion criteria All cases above 6 years presented with unilateral or bilateral ISSNHL Exclusion criteria Patient below 6 years old.

Data Collection

After fulfilling all inclusion and exclusion criteria all the patient will be subjected to:

* Full History taking including : the residency, occupation, duration of the clinical symptoms , associated symptoms like tinnitus , vertigo and aural fullness, the presence of previous episodes of hearing loss, the presence of any chronic medical condition especially diabetes and hypertension and neurological history, the medication history and surgical history specially ear surgeries, in addition to family history if relevant.
* Full medical examination including general examination with special emphasizing upon blood pressure measurements, full neurological examination, full ENT examination with vestibular testing especially in cases presented with vertigo
* Laboratory investigation Complete blood count test with differential to detect neutrophil lymphocyte monocyte ratio.

Renal function test Liver function test. Random blood sugar, oral glucose testing, HbA1c

audiological evaluation upon recruitment, all the patient will be subjected to audiological evaluation using audiogram where the hearing loss will be graded into mild, moderate, , sever and profound. speech discrimition will be graded into good ,fair and poor upon recruitment, all the patient will be subjected to audiological evaluation using ABR to asses retrocochlear pathology

Management plan

1. If the patient come at first two weeks of onset of hearing loss the patient will be manged by oral corticosteroid in the form of ,prednisolone60mg in two divided doses for 2 weeks.
2. Patient will be manged by 5 sessions of intratympanic steroid after failure of systemic steroid and patient who come after 2 weeks of onset of hearing loss , each session will be 3 days apart. The injectable material will be 1ml of hydrocortisone 8ml. The injection will be done under local anesthesia and microscope magnification. A pack of lidocaine gel will be applied in the external canal for 10 minutes in EAC to induce anesthesia by using insulin syringe 1ml bore.

An 8 ml of hydrocortisone will be injected in the ME through posteroinferior part of TM All patients will receive antiviral therapy in the form of acyclovir,valcyclovir All the patient will receive vasodilator.

Follow up All the patient will be subjected to audiological evaluation using the audiogram 2 weeks and one month after the initiation of the therapy to detect the treatment outcome.

Statistical analysis

* Factors affecting the treatment outcome will be grouped into

  1. Age.
  2. Onset of the disease.
  3. . tinnitus.
  4. vertigo.
  5. audiogram to detect the degree of hearing loss mild,moderate severe profund .speech discrimition low frequencies versus high frequencies.
  6. Complete blood count test with differential to detect neutrophil lymphocyte monocyte ratio.
  7. Comorbidities as hypertension cardiac All those factors will be compared to each other and to the final hearing outcome using correlation coefficient, regression analysis using the SPSS 20 software.

     Ethical consideration:

     . The Study will be reviewed by the Assiut University medical ethical committee as a study applied on humans to get their final approval.

     The aim of the study will be explained to each patient before the beginning of theprocess Written consent will be obtained from those who are willing to participate in thestudy.

     Privacy and confidentiality of all data will be assured .
* The aim of the study will be explained to each patient before the beginning of theprocess.

Written consent will be obtained from those who are willing to participate in the study.

Privacy and confidentiality of all data will be assured .

* Privacy and confidentiality of all data will be assured .
* . The Study will be reviewed by the Assiut University medical ethical committee as a study applied on humans to get their final approval.

The aim of the study will be explained to each patient before the beginning of theprocess Written consent will be obtained from those who are willing to participate in thestudy.

Privacy and confidentiality of all data will be assured .

• The aim of the study will be explained to each patient before the beginning of theprocess.

Written consent will be obtained from those who are willing to participate in the study.

Privacy and confidentiality of all data will be assured .

• Privacy and confidentiality of all data will be assured .

ELIGIBILITY:
Inclusion Criteria:

* All cases above 6 years presented with unilateral or bilateral ISSNHL

Exclusion Criteria:

* Patient below 6 years old

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
To detect if the duration between onset symptoms and start treatment ( in days) affect final hearing prognosis ( in decibel ) | 18months
  To detect if the duration between onset symptoms and start treatment ( in days) affect final hearing prognosis( in decibel) assessed by audiogram pre and post treatment
to detect if presence of comorbidities ( diabetes, hypertension, coronary heart diseases and chronic kidney disease ) affect the final hearing prognosis in decibel | 18months
  to detect if presence of comorbidities ( diabetes, hypertension, coronary heart diseases) from history taking affect the final hearing prognosis measured by decibel assessed by audiogram pre and post treatment
To detect if the severity of hearing loss symptoms in (decibel ) affect final hearing prognosis ( in decibel ) | 18 months
  To detect if the degree of hearing loss symptoms in (decibel) affect final hearing assessed by audiogram pre and post treatmentprognosis ( in s assessed by audiogram pre and post treatment
To detect if presence of associated presenting symptoms ( vertigo and tinnitus) affect the final hearing prognosis | 18 months
  To detect if presence of associated presenting symptoms ( vertigo and tinnitus) affect the final hearing prognosis ( in decibel) assessed by audiogram pre and post treatment

SECONDARY OUTCOMES:
To detect if the age in years affect the final hearing prognosis | 18 months
  To detect if the age in years affect the final hearing prognosis assessed by audiogram pre and post treatment
to detect if unilateral or bilateral symptoms affect the final hearing prognosis | 18 months
  to detect if unilateral or bilateral symptoms affect the final hearing prognosis assessed by pre and post treatment audiogram

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schreiber BE, Agrup C, Haskard DO, Luxon LM. Sudden sensorineural hearing loss. Lancet. 2010 Apr 3;375(9721):1203-11. doi: 10.1016/S0140-6736(09)62071-7. PMID 20362815
- [Result] Stachler RJ, Chandrasekhar SS, Archer SM, Rosenfeld RM, Schwartz SR, Barrs DM, Brown SR, Fife TD, Ford P, Ganiats TG, Hollingsworth DB, Lewandowski CA, Montano JJ, Saunders JE, Tucci DL, Valente M, Warren BE, Yaremchuk KL, Robertson PJ; American Academy of Otolaryngology-Head and Neck Surgery. Clinical practice guideline: sudden hearing loss. Otolaryngol Head Neck Surg. 2012 Mar;146(3 Suppl):S1-35. doi: 10.1177/0194599812436449. PMID 22383545
- [Result] Lin HC, Lee HC, Chao PZ, Wu CS. The effects of weather on the incidence of sudden sensorineural hearing loss: a 5-year population-based study. Audiol Neurootol. 2006;11(3):165-71. doi: 10.1159/000091268. Epub 2006 Feb 1. PMID 16462137
- [Result] Byl FM Jr. Sudden hearing loss: eight years' experience and suggested prognostic table. Laryngoscope. 1984 May;94(5 Pt 1):647-61. PMID 6325838
- [Result] Wei BP, Stathopoulos D, O'Leary S. Steroids for idiopathic sudden sensorineural hearing loss. Cochrane Database Syst Rev. 2013 Jul 2;2013(7):CD003998. doi: 10.1002/14651858.CD003998.pub3. PMID 23818120
- [Result] Trune DR, Canlon B. Corticosteroid therapy for hearing and balance disorders. Anat Rec (Hoboken). 2012 Nov;295(11):1928-43. doi: 10.1002/ar.22576. Epub 2012 Oct 8. PMID 23044978
- [Result] Lalaki P, Markou K, Tsalighopoulos MG, Daniilidis I. Transiently evoked otoacoustic emissions as a prognostic indicator in idiopathic sudden hearing loss. Scand Audiol Suppl. 2001;(52):141-5. doi: 10.1080/010503901300007344. PMID 11318448
- [Result] Han X, Yin X, Du X, Sun C. Combined Intratympanic and Systemic Use of Steroids as a First-Line Treatment for Sudden Sensorineural Hearing Loss: A Meta-Analysis of Randomized, Controlled Trials. Otol Neurotol. 2017 Apr;38(4):487-495. doi: 10.1097/MAO.0000000000001361. PMID 28207624
- [Result] Jung da J, Park JH, Jang JH, Lee KY. The efficacy of combination therapy for idiopathic sudden sensorineural hearing loss. Laryngoscope. 2016 Aug;126(8):1871-6. doi: 10.1002/lary.25751. Epub 2016 Mar 12. PMID 26972103
- [Result] Alexander TH, Harris JP. Incidence of sudden sensorineural hearing loss. Otol Neurotol. 2013 Dec;34(9):1586-9. doi: 10.1097/MAO.0000000000000222. PMID 24232060
- [Result] Arslan N, Oguz H, Demirci M, Safak MA, Islam A, Kaytez SK, Samim E. Combined intratympanic and systemic use of steroids for idiopathic sudden sensorineural hearing loss. Otol Neurotol. 2011 Apr;32(3):393-7. doi: 10.1097/MAO.0b013e318206fdfa. PMID 21221047
- [Result] Hu A, Parnes LS. Intratympanic steroids for inner ear disorders: a review. Audiol Neurootol. 2009;14(6):373-82. doi: 10.1159/000241894. Epub 2009 Nov 16. PMID 19923807